CLINICAL TRIAL: NCT03036137
Title: IMPACT OF TRANSCRANIAL DIRECT CURRENT STIMULATION ON THE STANDARDS OF CEREBRAL ELECTRIC ACTIVITY IN PATIENTS WITH CHRONIC TINNITUS: CLINICAL TRIAL, DOUBLE BLIND, PLACEBO-CONTROLLED
Brief Title: Impact of Neurostimulation on Patterns of Brain Electrical Activity in Patients With Tinnitus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Dayse da Silva Souza, Principal Investigator, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 61192416.9.0000.5188
Record Dates: First submitted 2017-01-25; First posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Tinnitus
Keywords: Tinnitus; Electroencephalogram; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Tinnitus | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Active Comparator): Subjects will receive 20 minutes of active tDCS for five consecutive days, current of 2 mA, in the temporoparietal left area, and right prefrontal cortex.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham tDCS (Sham Comparator): Subjects will receive 20 minutes of Sham tDCS for five consecutive days in the temporoparietal left area, and right prefrontal cortex.
  Interventions: Device: Sham Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Anodal stimulation of the temporoparietal left area with an cathode over the right dorsolateral prefrontal cortex. Stimulation will be applied for 20 minutes at 2 mA.
  Other Names: Direct current stimulator; Transcranial stimulator
  Arms: Active tDCS
Device: Sham Transcranial Direct Current Stimulation — Sham tDCS sessions will last 20 minutes
  Other Names: Sham stimulation
  Arms: Sham tDCS

SUMMARY:
Relating the electroencephalogram findings of patients with tinnitus before and after a therapeutic modality is still scarce in the literature, especially with neuromodulatory methods, more specifically with Transcranial Direct Current Stimulation - tDCS. This study is a double blind, sham-controlled clinical trial aiming investigate the impact of tDCS on patterns of brain electrical activity in patients with chronic tinnitus. 36 volunteers with tinnitus will be allocated randomly in 2 groups: the first (n = 18) will receive anodic tDCS in the temporoparietal left area and cathode in the right dorsolateral prefrontal cortex and the second group (n = 18) correspond to the sham group. In addition, healthy individuals (n = 18) will be recruited for comparative purposes of brain electrical activity with and without tinnitus, totaling 54 participants. Patients with tinnitus will receive transcranial direct current stimulation for 20 minutes for 5 consecutive days (1 week) and will be assessed before and after intervention by electroencephalogram, Acuphenometry, Visual Analogue Scale - VAS and questionnaire Tinnitus Handicap Inventory- THI. Follow-up of volunteers will also be performed after 1 month of the end of treatment with tDCS.

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 18 years;
* Chronic tinnitus for at least 6 months.
* Age-adjusted normal (sensorineural) hearing

Exclusion Criteria:

* Pregnancy and/or lactation;
* Concurrent treatment for tinnitus;
* Prior exposure to transcranial direct current stimulation (tDCS);
* History of epilepsy and/or seizures;
* Electronic implants or metallic objects in body;
* Skin conditions where electrodes will be applied;
* Major neurological co-morbidities.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2017-02-01 (Estimated); Primary Completion 2017-05-31 (Estimated); Study Completion 2017-09-01 (Estimated)

PRIMARY OUTCOMES:
Tinnitus Handicap Inventory | THI will be measured before intervention (baseline), after 5 daily sessions (day 5) and 1 month after the last intervention.
  Assesses change in tinnitus from baseline to follow-up periods post interventions

SECONDARY OUTCOMES:
Visual Analogue Scales (VAS) of perceived tinnitus loudness and distress | Visual analogue scale of tinnitus wiil be recorded at baseline (before intervention), before and after daily sessions with tDCS (day 1 to 5) , and 1 month after the last intervention.
  Self assessment of tinnitus loudness and tinnitus distress.
Acuphenometry | Acufhenometry wiil be recorded at baseline (before intervention), before and after daily sessions with tDCS (day 1 to 5) , and 1 month after the last intervention.
  Subjective assessment of the frequency, intensity and type of tinnitus.

CONTACTS AND LOCATIONS:
Locations (1):
- Dayse Souza, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: No